CLINICAL TRIAL: NCT05481801
Title: Adherence to Guidelines VAccination in Type 1 DIabetes Mellitus Patients (AVADI-2)
Acronym: AVADI-2
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: C-549
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — heterologous prime boost COVID-19 vaccination; Influenza Vaccines; Hepatitis B Vaccines; Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vaccination adherence: All type 1 diabetes adults patients attended in Ciudad Real General University Hospital willl be checked for Covid-19, Influenza Vaccination status, Pneumococcal Vaccination status and Hepatitis B Virus (HBV) status.
  Interventions: Biological: Covid-19 vaccination; Biological: Influenza vaccination; Biological: Pneumococal vaccination; Biological: Hepatitis B Virus (HBV) vaccination

INTERVENTIONS:
Biological: Covid-19 vaccination — Correct Covid19 vaccination status was considered in the following situation:
  Received at least two Covid-19 vaccine doses being the last in the last 6 months.
Biological: Influenza vaccination — Correct influenza vaccination status was considered in the following situation:
  - Received at least one Influenza vaccine dose in the last year.
Biological: Pneumococal vaccination — Correct pneumococal vaccination status was considered if a subject received at least one of the following options:
  One pneumococcal conjugate vaccine (PCV) 13 dose in the last year. One PCV13 dose following a pneumococcal polysaccharide vaccine (PPSV) 23 dose between the following 8 weeks and 12 months.
  One PPSV 23 dose in the last 5 years. One PPSV23 dose in the last 5 years and a second PPSV23 dose at 5 years or PCV13 at 1 year.
Biological: Hepatitis B Virus (HBV) vaccination — Correct Hepatitis B Virus (HBV) vaccination status was considered in the following situation:
  .- Received at least three consecutive doses of HBV vaccine during six consecutive months.

SUMMARY:
Observational study about adherence to guidelines for Covid-19, Influenza, Pneumococcal and Hepatitis B Vaccination in adult patients with type 1 Diabetes mellitus.

DETAILED DESCRIPTION:
Cross-sectional analysis about adherence to guidelines for Covid-19, Influenza, Pneumococcal and Hepatitis B Vaccination in adult patients with type 1 Diabetes mellitus.

All clinical variables are gathered from two EMR softwares (Mambrino XXI and Turriano).

Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee. All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age: 18 yrs. or older

Exclusion Criteria:

* Other diabetes types.
* Younger than 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All type 1 diabetes patients attendet at the Ciudad Real General University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Vaccination adherence | 1 year and a half
  Adherence ratio (number of vaccinated patients/total number of patients) to regional guidelines for the Immunization for Covid-19, pneumococcus, influenza and HBV of Adults With Type 1 Diabetes Mellitus

SECONDARY OUTCOMES:
Sick Leaves | 1 year and a half
  Total number of related sick leaves due to Covid-19, pneumococcus, influenzae or HBV according to vaccination status (vaccinated or not vaccinated).
Hospital admission | 1 year and a half
  Number of hospital admission according to vaccination status (vaccinated or not vaccinated) for Covid-19, pneumococcus, influenza and HBV.
Death | 1 year and a half
  Mortality rate according to vaccination status

CONTACTS AND LOCATIONS:
Locations (1):
- Ciudad Real General University Hospital, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: No
Clinical IPD will be available at request from others researchers.

REFERENCES:
- [Result] Moreno-Fernandez J, Garcia-Seco JA, Rodrigo EMO, Segura AMS, Garcia-Seco F, Munoz-Rodriguez JR. Vaccination adherence to influenza, pneumococcal and hepatitis B virus in adult type 1 diabetes mellitus patients. Prim Care Diabetes. 2020 Aug;14(4):343-348. doi: 10.1016/j.pcd.2019.09.004. Epub 2019 Sep 30. PMID 31582202
- [Result] Giatraki V, Dimitriou H, Pappas A, Mamoulakis D, Makris G, Galanakis E, Perdikogianni C. Vaccine coverage in children, adolescents and adults with type 1 diabetes and their close contacts in Crete. Hum Vaccin Immunother. 2021 Nov 2;17(11):4291-4298. doi: 10.1080/21645515.2021.1973882. Epub 2021 Oct 6. PMID 34613871
- [Result] Wang CH, Jones J, Hilliard ME, Tully C, Monaghan M, Marks BE, Hildebrandt T, Streisand R. Correlates and Patterns of COVID-19 Vaccination Intentions among Parents of Children with Type 1 Diabetes. J Pediatr Psychol. 2022 Aug 12;47(8):883-891. doi: 10.1093/jpepsy/jsac048. PMID 35689648